CLINICAL TRIAL: NCT04928508
Title: Phase 1 Trial of OK-1 (SHetA2) in Patients With Advanced or Recurrent Solid Tumors
Brief Title: Advanced or Recurrent Solid Tumors Treated With SHetA2
Acronym: Okgyn1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OU-SCC-OKGyn1; R01CA196200 (NIH)
Record Dates: First submitted 2021-06-10; First posted 2021-06-16 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OK-1 capsule (Experimental): OK-1 (oral, BID) within a 21-days cycle
  Interventions: Drug: OK-1

INTERVENTIONS:
Drug: OK-1 — OK-1 orally in the form of 50 mg capsules. Four dose levels will be evaluated:
  5.4mg/kg 7.0mg/kg 9.0mg/kg 12mg/kg
  Other Names: NSC 726189

SUMMARY:
The purpose of this research is to test the safety of the study drug (OK-1) and see what effects (good and bad) this drug has on patients with recurrent solid tumors.

DETAILED DESCRIPTION:
OK-1 capsules will be given twice a day, every day in 21-day blocks of time. Each block of time is called a cycle. The cycle will be repeated until the patient or doctor no longer feel participation in the study is right for the patient. There will be lab tests and examinations to monitor the patients progress. We expect that taking part in this research will last up to three years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic diagnosis of recurrent solid tumor which has progressed through available therapies with expected survival benefit. Histologic documentation of the original primary tumor is required via the pathology report.

Patients must have adequate:

* Bone marrow function as defined per protocol
* Renal function as defined per protocol
* Hepatic function as defined per protocol
* International normalized ratio (INR) or prothrombin time (PT) ≤1.5x ULN unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) ≤1.5x ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Neurologic function: Neuropathy (sensory and motor) less than or equal to Grade 1. Patients should be free of active infection requiring parenteral antibiotics or a serious uncontrolled medical illness or disorder within four weeks of study entry.
* Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration. Continuation of hormone replacement therapy is permitted.
* Patients must have a performance status score of 0-2 by Eastern Cooperative Group (ECOG) criteria.
* Patients of childbearing potential must have a negative pregnancy test prior to the study entry and be practicing an effective form of contraception. If applicable, patients must discontinue breastfeeding prior to study entry.
* Patients must have satisfactory results for the baseline laboratory analyses and diagnostic procedures as specified in the protocol
* Patients must have signed an IRB-approved informed consent and authorization permitting release of personal health information.
* Patients must be at least 18 years old.
* Patients in all cohorts must have a fresh pre-treatment tumor biopsy. This is optional only for patients enrolled on dose level 2 and 3. Biopsies are mandatory on cohort 4 and/or expansion.
* Patients must be willing to have fresh biopsy taken post-Cycle 1 treatment (optional only for patients enrolled on dose level 2 and 3; Biopsies are mandatory for patients enrolling on Cohort 4 and/or dose expansion phase.)
* Life expectancy of at least 3 months.
* Patients must be able to take oral medications.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

Exclusion Criteria:

* Unable to take oral medications
* Patients of childbearing potential not practicing adequate contraception, patients who are pregnant, or patients who are breastfeeding are not eligible for this trial
* Patients who are pregnant or breastfeeding or expecting to conceive children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to OK-1.
* A diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Patients receiving treatment for active autoimmune disease. "Active" refers to any condition currently requiring therapy. Examples of autoimmune disease include systemic lupus erythematosus, multiple sclerosis, inflammatory bowel disease and rheumatoid arthritis. (note if steroid use is <10mg/day prednisolone equivalent and patient has stable symptoms they may be allowed on study with discussion with the medical monitor)
* Patients with a prior or concurrent malignancy whose natural history or treatment does have the potential to interfere with the safety or efficacy assessment of the investigational regimen are NOT eligible for this trial.
* Known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus ribonucleic acid [HCV RNA] [qualitative] is detected). Ongoing systemic bacterial, fungal, or viral infection; known human immunodeficiency virus (HIV) infection with positive viral load or acquired immunodeficiency syndrome (AIDS)-related illness. Patients with HIV and a negative viral load are allowed on study.
* Patients with concurrent severe medical problems unrelated to the malignancy that would significantly limit full compliance with the study or expose the patient to extreme risk or decreased life expectancy.
* Patients with history or evidence upon physical examination of CNS disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of treatment on this study.

NOTE: Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging (using the identical imaging modality for each assessment, either magnetic resonance imaging [MRI] or computed tomography [CT] scan) for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. Carcinomatous meningitis precludes a patient from study participation regardless of clinical stability

* Patients taking concomitant therapy with any of the following: other non-study cytotoxic chemotherapy; other investigational therapies.
* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Prior chemotherapy or targeted small molecule therapy within 4 weeks, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

Note: Patients with ≤ Grade 2 neuropathy or ≤ Grade 2 alopecia are an exception to this criterion and may qualify for the study.

Note: If the patient underwent major surgery, she must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.

* Prior bone marrow/hematopoietic stem cell transplantation
* History of solid organ, bone marrow, or progenitor cell transplantation
* History of major surgical procedure within 28 days prior to start of study treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of dose-limiting toxicities of treatment with OK-1 | 21 days
Dosage Recommendation for Phase 2 | 21 days

SECONDARY OUTCOMES:
Rate of objective response | up to three years
Median duration of response | up to three years
Rate of disease control | up to three years
Median progression free survival | up to three years
Median overall survival | up to three years
Incidence of adverse events | up to three years
  safety and tolerability of OK-1 using Common Terminology Criteria for Adverse Events (CTCAE) v.5.0
Tmax of PK plasma concentration | 24 hours
Cmax of PK plasma concentration | 24 hours
AUC of PK plasma concentration | 24 hours
t1/2 of PK plasma concentration | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Debra Richardson, MD, Principal Investigator — Stephenson Cancer Center
Locations (1):
- Stephenson Cancer Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No